CLINICAL TRIAL: NCT05601505
Title: Circulating Tumor DNA-guided Neoadjuvant Treatment Strategy for Locally Advanced Rectal Cancer --- a Multicenter Randomized Controlled Trial (CINTS-R)
Brief Title: Circulating Tumor DNA-guided Neoadjuvant Treatment Strategy for Locally Advanced Rectal Cancer
Acronym: CINTS-R
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-PUMCH-C-005
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced Rectal Carcinoma; Circulating Tumor DNA
Keywords: Locally advanced rectal cancer; circulating tumor DNA; Neoadjuvant chemoradiotherapy; Total neoadjuvant therapy; Randomized Controlled Trial
MeSH Terms: interventions — Circulating Tumor DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional neoadjuvant chemoradiotherapy group (No Intervention): Eligible patients randomized into arm A will receive traditional neoadjuvant chemoradiotherapy, including long-course radiotherapy with a total number of 45-50.4Gy in 25-28 fractions, and with concurrent 3 times of oral capecitabine, the strategies of capecitabine are:
  During radiotherapy: capecitabine 1650mg/m2/d, orally administered twice a day, d1-d14, every 3 weeks as a course; During the non-radiotherapy period: capecitabine 2000mg/m2/d, orally administered twice daily, d1-d14, every 3 weeks as a course
- ctDNA-guided neoadjuvant treatment group (Experimental): After sequencing tumor tissue, those with MSI-H/TMB-H or POLD/POLE2 mutation willed be arranged to receive immune therapy following NCRT，Terelizumab，200mg.
  The others are arranged to randomly receive TNT (VAF>0.4%) or NCRT (VAF<0.4%) according to VAF value by the level of ctDNA.
  TNT： Long course radiotherapy combined with 2 courses of single-agent capecitabine chemotherapy → 6 courses of CapeOX (Capecitabine 2000mg/m2/ day, twice orally, d1-14; Oxaliplatin 100-130mg/m2, intravenous infusion, d1; Every 3 weeks for a course of treatment.) chemotherapy was performed 2 to 3 weeks after the end of chemotherapy.
  Interventions: Other: circulating tumor DNA

INTERVENTIONS:
Other: circulating tumor DNA — This study will further testify the prognostic value of ctDNA in the treatment term of locally advanced rectal cancer, the higher the VAF value, the higher the risk of recurrence and metastasis.
  Arms: ctDNA-guided neoadjuvant treatment group

SUMMARY:
Rectal cancer still remains one of the most popular tumors, however, distance metastasis still remains as high as 30% and the long-term survival outcomes are still unsatisfying. The recent conception of total neoadjuvant therapy and immune therapy is becoming popular and the oncologic effects are encouraging, especially in terms of circulating tumor DNA (ctDNA), the prognostic value of ctDNA has been demonstrated by our prior study. This study will carry out accurate ctDNA-guided neoadjuvant therapy on the basis of previous studies of the research group, and give appropriate treatment plans and treatment intensity to patients with different disease degrees. At the same time, combined with the latest progress in clinical diagnosis and treatment, the potential beneficiaries of immunotherapy were screened scientifically, and the combined immunotherapy was implemented accordingly.

DETAILED DESCRIPTION:
Rectal cancer still remains one of the most popular tumors, a multidisciplinary approach including neoadjuvant chemoradiotherapy, total mesorectal excision and adjuvant chemotherapy has resulted a satisfying oncologic outcome in terms of reducing local recurrence and improving local control of disease for the treatment of rectal cancer, however, distance metastasis still remains as high as 30% and the long-term survival outcomes is still unsatisfying.

The recent conception of total neoadjuvant therapy and immune therapy is becoming popular and the oncologic effects are encouraging, especially in terms of circulating tumor DNA (ctDNA), the prognostic value of ctDNA has been demonstrated by our prior study. This study demonstrated that ctDNA is an effective marker of tumor burden in real time and for the first time identified baseline ctDNA mutation frequency before nCRT as an independent prognostic factor for recent LARC recurrence and metastasis. This suggests that patients with different tumor burden according to baseline ctDNA mutation frequency should be given neoadjuvant therapy with corresponding intensity, in order to improve systemic disease control in patients with high risk of recurrence and metastasis, and to avoid overtreatment in patients with low risk.

In conclusion, this study will carry out accurate ctDNA-guided neoadjuvant therapy on the basis of previous studies of the research group, and give appropriate treatment plans and treatment intensity to patients with different disease degrees. At the same time, combined with the latest progress in clinical diagnosis and treatment, the potential beneficiaries of immunotherapy were screened scientifically, and the combined immunotherapy was implemented accordingly. With the development of this study, several precision medicine research results obtained by our research group will be expected to be translated into clinical practice as soon as possible, which will improve the efficacy of LARC patients, reduce the rate of adverse reactions, and ultimately promote the improvement of the treatment level of rectal cancer and the more reasonable use of public medical resources.

The patients with locally advanced rectal cancer staged as cT3-4N0/cTanyN+ will be included in this study. Patients will be randomized into two groups, the experimental group will receive different strategies after next generation sequencing of tumor tissue and IMC, those with MSI-H or TMB-H will be advised to receive immune therapy, and the others will be arranged to randomly receive NCRT (baseline VAF<0.5%) or total neoadjuvant therapy (TNT) (baseline VAF≥0.5% or a positive post-CRT ctDNA) according to the VAF value of ctDNA; the control group will receive modified NCRT only.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years;
2. ECOG score 0-2;
3. Rectal adenocarcinoma confirmed by pathology;
4. The lower margin of the tumor was less than 12cm from the anal margin;
5. Patients with clinical stage cT3-4N0M0 or cTanyN+M0;
6. Newly treated patients who have not received treatment including radiotherapy, chemotherapy and surgery;
7. Liver, kidney and other organs have good function and can tolerate radiotherapy, chemotherapy and surgery;
8. Patients and family members can understand the study protocol, voluntarily participate in the study and sign informed consent.

Exclusion Criteria:

1. ECOG score > 2;
2. Patients with multiple primary colorectal cancers;
3. A history of other malignant tumors (other than cured basal cell carcinoma, cervical carcinoma in situ, surgically treated localized prostate cancer, or surgically resected breast ductal carcinoma in situ) within the past 5 years;
4. Complicated with intestinal obstruction, intestinal perforation, gastrointestinal bleeding and other patients requiring emergency surgery;
5. pregnant or lactating women;
6. Patients with a history of severe mental illness, immune disease, hormone medication;
7. Patients contraindicated by MRI examination, chemoradiotherapy, immunotherapy or surgery;
8. Participated in other clinical researchers in the past 3 months;
9. Any other circumstances that the investigator considers inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
two-year disease-related treatment failure, 2y-DrTF | 2 years
  the incidence of any of the following events occurring after treatment: identification of distant metastasis or progression to unresectable disease before surgery, non-radical resection of the primary tumour, local recurrence or distant metastasis after radical surgery, new primary colorectal tumour, or treatment-related death.

SECONDARY OUTCOMES:
Time to recurrence, TTR | 2 years
  The median time from randomization to the first observation of recurrence.
Two-year overall survival, 2yOS | 2 years
  Refers to the proportion of patients still alive at 2 years after surgery
two-year disease-free survival (2yDFS) | 2 years
  the percentage of patients who remain free of cancer recurrence or death from any cause two years after surgery.
clinical complete response (cCR) and near complete response (ncCR) rate | up to 1 year
  cCR and ncCR rate evaluated based on comprehensive examinations according to NCCN guidelines.
pathologically complete response (pCR) rate | up to 1 year
  the percentage of patients who are assessed as pathologically complete response (pCR) by pathologist.
pathological tumour regression grade (pTRG) | up to 1 year
  pathological tumor regression grade which is determined according to the criteria of the American Joint Committee on Cancer (AJCC) 8th edition
Quality of life assessment (QoL) | 5 years
  it will be assessed by European Organization for Research and Treatment of Cancer (EORTC) questionnaires at each follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Peking Union Medical College Hospital, Peking Union Medical College and Chinese Academy of Medical Sciences,, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript will be available from the corresponding author at reasonable request. They may only be shared under the terms of a Data Use Agreement. Data from this clinical trial will only be shared in compliance with national regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The datasets analyzed during the current study and other supporting information will be available no earlier than 1 year following the date of publication.
Access Criteria: IPD and supporting information can be accessed based on reasonable request by contacting the corresponding author.

REFERENCES:
- [Derived] Zhang X, Zhou J, Geng J, Li Y, Huang F, Shu W, Fu W, Zhou X, Wu G, Jia W, Cui J, Wang Z, Han J, Shi B, Li L, Rui J, Xue H, Hu K, Xu T, Chen W, Lu J, Yao H, Liu Q, Lin G. Feasibility of ctDNA-guided precision neoadjuvant therapy in locally advanced rectal cancer: Insights from the ongoing CINTS-R trial. Eur J Cancer. 2026 Feb 5;234:116193. doi: 10.1016/j.ejca.2025.116193. Epub 2025 Dec 18. PMID 41435753
- [Derived] Zhou J, Zhang X, Liu Q, Li Y, Wu G, Fu W, Yao H, Wang Z, Xue H, Xu T, Chen W, Lu J, Zhang G, Wu B, An Y, Qiu X, Xiao Y, Lin G. Rationale and design of a multicentre randomised controlled trial on circulating tumour DNA-guided neoadjuvant treatment strategy for locally advanced rectal cancer (CINTS-R). BMJ Open. 2025 Feb 2;15(1):e090765. doi: 10.1136/bmjopen-2024-090765. PMID 39894522